CLINICAL TRIAL: NCT02976545
Title: VECU EMOTIONNEL CHEZ LES PATIENTES SOUFFRANT DE CRISES NON EPILEPTIQUES PSYCHOGENES : ETUDE EN IMAGERIE PAR RESONANCE MAGNETIQUE FONCTIONNELLE-ETUDE EMOCRISES
Brief Title: Emotional Lived in Patients Suffering From Psychogenic Nonepileptic Seizures : Study by Functional Magnetic Resonance Imaging
Acronym: EMOCRISES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, M.D. Coraline HINGRAY, Doctor, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-A01295-46
Record Dates: First submitted 2016-11-25; First posted 2016-11-29 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Psychogenic Non-epileptic Seizures
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNES (Other): Psychogenic Non-epileptic Seizures subjects
  Interventions: Device: fMRI (functional Magnetic Resonance Imaging); Behavioral: psychiatric evaluation
- PTSD (Other): Post Traumatic Stress Disorder
  Interventions: Device: fMRI (functional Magnetic Resonance Imaging); Behavioral: psychiatric evaluation
- Healthy controls (Other): Healthy controls
  Interventions: Device: fMRI (functional Magnetic Resonance Imaging); Behavioral: psychiatric evaluation

INTERVENTIONS:
Device: fMRI (functional Magnetic Resonance Imaging) — fMRI examination
Behavioral: psychiatric evaluation — psychiatric evaluation

SUMMARY:
Currently, hypothetical models of understanding Psychogenic Non-epileptic Seizures (PNES) involve emotional dysregulation.

The hypothesis of a disorder of emotional experience is mainly based on behavioral data and disturbance of autonomic responses in response to images in emotional content (Mignot et al 2015, in submission; Bakvis et al 2013). Various imaging studies have identified brain structures belonging to the limbic system in particular that seem functionally impaired in this population. These functional connectivity abnormalities are correlated with dissociation scores in PNES patients (Van der Kruijs et al 2012 and 2014).

Investigators propose to specifically study the brain activity of PNES patients during tasks emotional content to identify the mechanisms involved in this emotional dysregulation. This work is essential to understanding the mechanisms and the development of new therapeutic strategies

ELIGIBILITY:
Common Inclusion Criteria:

* Female,
* Right-handed
* Affiliation to the French social security system,
* Informed signing of the study consent.

Specific Inclusion Criteria for PNES group :

* PNES diagnosed by a neurologist specialized in epilepsy, based on clinical symptoms analysis and video-EEG recording,
* Absence of concomitant epilepsy.

Specific Inclusion Criteria for PTSD group : PTSD diagnosed by a psychiatrist, based on clinical symptoms as recorded in DSM5 (Diagnostic and Statistical Manual of Mental Disorders).

Specific Inclusion Criteria for healthy controls : Healthy controls will be paired up with patients on age and level of schooling criteria.

Exclusion Criteria:

common criteria for all groups:

* Neurological history or comorbidity (epilepsy included),
* Current neurological treatment,
* Posology change or introduction of psychoactive treatment dating back to less than a month,
* Psychotic comorbidity (schizophrenia),
* Addiction history apart for smoking,
* History of head trauma,
* Mental retardation,
* Being the subject of articles L.1121-5 to L.1121-8 and L1122-1-2 of the French Code of Public Health (i.e. being a not responsible adult),
* Lack of French language proficiency or inability to understand instructions,
* Uncorrected visual impairment,
* Any contraindication to MRI (pacemaker, ferromagnetic foreign body, claustrophobia, etc.).

Specific exclusion Criteria for PNES group : Diagnosis of PNES challenged or denied by the patient.

Specific exclusion Criteria for PTSD group :

* Diagnosis of PTSD challenged or denied by the patient, current or history of functional neurological symptom disorder,
* History of PNES (conversion disorder).

Specific exclusion Criteria for healthy controls :

* History of PTSD,
* History of PNES (conversion disorder).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Brain activity | 6 months after the last inclusion
  To compare brain activity during emotional tasks in fMRI (Blood-Oxygen-Level-Dependent contrast sequences) between: patients suffering from PNES, patients suffering from PTSD and healthy controls, with age and education level matching.

SECONDARY OUTCOMES:
Valence and intensity of the emotional images | 6 months after the last inclusion
  To compare subjective experience rating across the three groups, during emotional pictures watching task;
Cerebral functional connectivity | 6 months after the last inclusion
  To compare differences of cerebral functional connectivity (main physiological brain networks) in resting state fMRI across the tree groups
"Dissociative Experience Scale (DES) questionnaire" score and "Toronto Alexithymia Scale (TAS20) questionnaire" score | 6 months after the last inclusion
  To study the correlation between cerebral activity and level of dissociation (DES) and alexithymia (TAS20) in PNES and PTSD groups

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France

REFERENCES:
- [Background] Fauve P, Tyvaert L, Husson C, Hologne E, Gao X, Maillard L, Schwan R, Banasiak C, El-Hage W, Hossu G, Hingray C. Functional MRI-based study of emotional experience in patients with psychogenic non-epileptic seizures: Protocol for an observational case-control study-EMOCRISES study. PLoS One. 2022 Jan 7;17(1):e0262216. doi: 10.1371/journal.pone.0262216. eCollection 2022. PMID 34995332